CLINICAL TRIAL: NCT03932682
Title: A Phase 3, Randomized, Observer-blind, Multicenter Study to Evaluate the Efficacy, Immunogenicity and Safety of Seqirus' Cell-Based Quadrivalent Subunit Influenza Virus Vaccine (QIVc) Compared to a Non-Influenza Vaccine When Administrated in Healthy Subjects Aged 6 Months Through 47 Months
Brief Title: Efficacy Study With QIVc in Pediatric Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V130_14; 2018-001857-29 (EudraCT Number)
Record Dates: First submitted 2019-04-22; First posted 2019-05-01 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Influenza, Human
Keywords: Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial is designed as an observer-blind study. During the treatment period of the study, only designated, trained unblinded personnel will be responsible for administering the study vaccines to the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- QIVc (Experimental): Cell-derived Quadrivalent Influenza Vaccine
  Interventions: Biological: QIVc
- Comparator (Active Comparator): Non-influenza Comparator
  Interventions: Biological: Comparator

INTERVENTIONS:
Biological: QIVc — QIVc is a quadrivalent vaccine and contains 2 influenza type A strains and 2 influenza type B lineages recommended by World Health Organization (WHO) for inclusion in the quadrivalent vaccine formulation for the influenza season corresponding to the season of conduct of study.
  Other Names: Flucelvax Quadrivalent
  Arms: QIVc
Biological: Comparator — Meningococcal Group C Polysaccharide Conjugate Vaccine (NeisVac-C)
  Arms: Comparator

SUMMARY:
This phase 3 clinical study is a randomized, observer-blind, multicenter study of QIVc versus a non-influenza vaccine in subjects 6 months though 47 months of age. The purpose of this study is to evaluate efficacy of QIVc in the prevention of laboratory confirmed influenza A or B disease in children 6 through 47 months of age, compared to a non-influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, all subjects must meet all of the inclusion criteria described.

* Individuals of 6 through 47 months of age on the day of informed consent.
* Individuals whose parent(s)/Legally Acceptable Representative (LAR) have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
* Individuals who can comply with study procedures including follow-up.
* Individuals in generally good health as per the Investigator's medical judgement.

If applicable, prior to receipt of second study vaccination, subjects must be evaluated to confirm that they are eligible for subsequent vaccination. If subjects do not meet the criteria of the original inclusion criteria listed above, they should not receive additional vaccinations.

Exclusion Criteria:

* Acute (severe) febrile illness. Enrollment could be considered if the fever is absent for 72 hours.
* History of any anaphylaxis, serious vaccine reactions or hypersensitivity, including allergic reactions, to any component of vaccine or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws. These may include known bleeding disorders, or treatment with anticoagulants in the 3 weeks preceding vaccination.
* A known history of Guillain-Barré Syndrome or other demyelinating diseases such as encephalomyelitis and transverse myelitis.
* Abnormal function of the immune system resulting from a clinical condition
* Received influenza vaccination or has had documented influenza disease in the last 6 months prior to informed consent.
* Prior vaccination to prevent Neisseria meningitides serogroup C disease or prior infection caused by this organism.

Additional eligibility criteria are provided in the study protocol.

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5723 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (74):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh
- Bulgaria (7):
  - 10008-Medical Center Viva Feniks, Dobrich
  - 10007-MHAT Dr. Stamen Iliev AD, Montana
  - 10003-UMHAT Dr. Georgi Stranski EAD, Pleven
  - 10002-UMHAT Sveti Georgi EAD, Plovdiv
  - 10006-UMHAT-Plovdiv AD, Plovdiv
  - 10004-SHATPPD Dr Dimitar Gramatikov Ruse EOOD, Rousse
  - 10009-Medical Center Unimed Eood, Sevlievo
- Czechia (5):
  - 20303-MUDr. Stefan Hrunka, Prakticky lekar pro deti a dorost, Chlumec nad Cidlinou
  - 20301-MUDr. Daniel Drazan, Prakticky lekar pro deti a dorost, Jindřichův Hradec
  - 20302-MUDr. Daniela Pniakova s.r.o., Ostrava
  - 20304-MUDr. David Zeman s.r.o., Ostrava-poruba
  - 20305-MUDr. Iva Madejova, Prakticky lekar pro deti a dorost, Pardubice
- Estonia (6):
  - 23305-Vee Family Doctor's Centre, Paide
  - 23301-Innomedica OÜ, Tallinn
  - 23303-Al Mare Perearstikeskus OU, Tallinn
  - 23304-Merelahe Family Doctors Center, Tallinn
  - 23307-Tallinn Children's Hospital, Tallinn
  - 23302-Clinical Research Centre, Tartu
- Honduras (3):
  - 34001-Demedica, San Pedro Sula
  - 34003-Clínica Médica y Dental CLIMEDENTY, Tegucigalpa
  - 34002-Inversiones en Investigación Médica (INVERIME), Tegucigalpa
- 42802-OLVI Medical Centre, Daugavpils, Latvia
- Malaysia (5):
  - 45804-Clinical Research Centre (CRC), Hospital Tuanku Fauziah, Kangar, Perlis
  - 45803-Sarawak General Hospital, Kuching, Sarawak
  - 45802-Hospital Sibu, Sibu, Sarawak
  - 45805-Klinik Kesihatan Putrajaya Presint 9, Putrajaya, Wilyah Persekutuan Putrajaya
  - 45801-University Malaya Medical Centre, Kuala Lumpur
- New Zealand (2):
  - 55403-Christchurch Clinical Studies Trust, Christchurch
  - 55401-Wellington Hospital, Wellington
- Pakistan (5):
  - 58602-Shifa International Hospital, Islamabad
  - 58604-The Aga Khan, Karachi
  - 58605-Avicenna Hospital, Lahore
  - 58607-Central Park Teaching Hospital, Lahore
  - 58601-Al Shifa Research Centre, Rawalpindi
- Philippines (12):
  - 60808-University of the Philippines Manila Development Foundation Inc, Ermita, Manila
  - 60810-UERM Memorial Medical Center, Quezon City, Quezon
  - 60817-Health Index Multispecialty Clinic, Bacoor
  - 60801-Chong Hua Hospital, Cebu City
  - 60812-De La Salle Medical and Health Sciences Institute, Dasmariñas
  - 60816-De La Salle Medical and Health Sciences Institute, Dasmariñas
  - 60806-Mary Chiles General Hospital, Manila
  - 60814-Philippine General Hospital, Manila
  - 60815-Philippine General Hospital, Manila
  - 60818-Philippine General Hospital, Manila
  - 60811-UERM Memorial Medical Center, Quezon City
  - 60813-Philippine Children's Medical Center, Quezon City
- Poland (8):
  - 61605-Osrodek Badan Klinicznych IN-VIVO sp. z o.o., Bydgoszcz
  - 61603-Jerzy Brzostek Prywatny Gabinet Lekarski, Dębica
  - 61607-Gdanskie Centrum Zdrowia Sp. z o.o., Gdansk
  - 61604-Hanna Czajka, Indywidualna Specjalistyczna Praktyka Lekarska, Krakow
  - 61608-Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - 61602-Niepubliczny Zaklad Lecznictwa Ambulatoryjnego Michalkowice, Siemianowice Śląskie
  - 61601-ETG Network- Skierniewice,Clinmed Research, Skierniewice
  - 61609-Szpital im. Swietej Jadwigi Slaskiej w Trzebnicy, Trzebnica
- Romania (4):
  - 64201-SC Sana Monitoring SRL., Bucharest
  - 64202-Spitalul Municipal Caracal, Caracal
  - 64205-Sc Med Fam Apolo srl, Călăraşi
  - 64206-S.C Centrul Clinic Mediquest S.R.L, Sângeorgiu de Mureş
- South Africa (9):
  - 71006-Madibeng Centre for Research, Brits
  - 71004-Tread Research, Cape Town
  - 71007-Allergy & Immunology Unit, Cape Town
  - 71002-Synergy Biomed Research Institute, East London
  - 71009-Perinatal HIV Research Unit, Tshepong Hospital, Klerksdorp
  - 71001-Be Part Yoluntu Centre, Paarl
  - 71008-Clinical Trial Systems, Pretoria
  - 71003-Soweto Clinical Trials Centre, Soweto
  - 71005-Limpopo Clinical Research Initiative, Thabazimbi
- Thailand (3):
  - 76405-Phramongkutklao Hospital, Ratchathewi, Bangkok
  - 76401-Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok
  - 76404-Department of Tropical Pediatrics, Faculty of Tropical Medicine, Mahidol University, Bangkok
- Ukraine (3):
  - 80404-Reg Mun NPE Chernivtsi RCCH Infectious Dept for Infants SHEI of UBSMU, Chernivtsi
  - 80405-CI Dnipro Children's City CH #5 of Dnipro City Council, Dnipro
  - 80401-Vinnytsia RCCH Policlinic Dept Vinnytsia M.I.Pyrogov NMU, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Seqirus will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact Seqirus at seqirus.clinicaltrials@seqirus.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment period: Previously vaccinated subjects: Day of vaccination to 28 days after vaccination (Day 1-Day 29); Not previously vaccinated subjects: Day of first vaccination to 28 days after second vaccination (Day 1-Day 57) Study completion: At end of influenza season and at least 180 days after last vaccination during treatment period, whichever was longer (previously vaccinated subjects: Day 181/end of influenza season; not previously vaccinated subjects: Day 209/end of influenza season)
Period: Overall Study
Arm/Group | QIVc | Comparator
Started (QIVc Arm: Previously vaccinated subjects: 1 dose QIVc. Not previously vaccinated subjects: 2 doses (QIVc/QIVc) during treatment period; all subjects aged 6 through 11 months at enrollment received 1 dose of NeisVac-C at study completion. Comparator Arm: Previously vaccinated subjects: 1 dose NeisVac-C. Not previously vaccinated subjects: 2 doses (NeisVac-C/Placebo) during treatment period; all subjects aged 6 through 11 months at enrollment received 1 dose of NeisVac-C at study completion.) | 2860 | 2863
Completed | 2794 | 2766
Not Completed | 66 | 97
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 37 | 45
Not completed — Lost to Follow-up | 19 | 25
Not completed — Protocol Violation | 0 | 2
Not completed — Other | 9 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QIVc | Comparator | Total
Number analyzed (Participants) | 2860 | 2863 | 5723
Age, Continuous [Mean (Standard Deviation); unit: months] | 25.8 (11.9) | 25.9 (11.9) | 25.9 (11.9)
Age, Customized [Count of Participants; unit: Participants]
  6 months through 23 months | 1268 | 1264 | 2532
  24 months through 47 months | 1592 | 1599 | 3191
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1418 | 1333 | 2751
  Male | 1442 | 1530 | 2972
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 155 | 157 | 312
  Not Hispanic or Latino | 2696 | 2697 | 5393
  Unknown or Not Reported | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1098 | 1096 | 2194
  Black or African American | 348 | 349 | 697
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 1239 | 1234 | 2473
  Other | 175 | 183 | 358
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 38 | 33 | 71
  Czechia | 41 | 38 | 79
  Philippines | 608 | 609 | 1217
  Ukraine | 184 | 183 | 367
  Malaysia | 31 | 34 | 65
  Thailand | 72 | 69 | 141
  New Zealand | 7 | 7 | 14
  Bangladesh | 101 | 99 | 200
  Latvia | 3 | 2 | 5
  Pakistan | 279 | 282 | 561
  Poland | 217 | 220 | 437
  Honduras | 147 | 151 | 298
  South Africa | 376 | 380 | 756
  Bulgaria | 131 | 135 | 266
  Estonia | 625 | 621 | 1246
Previous influenza vaccination [Count of Participants; unit: Participants]
  Previously vaccinated | 48 | 62 | 110
  Not previously vaccinated | 2812 | 2801 | 5613
Participants enrolled in each influenza season [Count of Participants; unit: Participants] — Season 1 = Southern Hemisphere (SH) 2019; Season 2 = Northern Hemisphere (NH) 2019/2020; Season 3 = NH 2020/2021; Season 4 = NH 2022/2023; Season 5 = SH 2023.
  Participants
    Season 1 | 344 | 349 | 693
    Season 2 | 497 | 489 | 986
    Season 3 | 525 | 521 | 1046
    Season 4 | 496 | 504 | 1000
    Season 5 | 998 | 1000 | 1998
Body mass index [Mean (Standard Deviation); unit: kg/m2] — Population: Two subjects (one subject in each vaccine group) did not have body mass index data.
  kg/m2
    number analyzed (Participants) | 2859 | 2862 | 5721
    (all) | 16.51 (2.2) | 16.61 (2.9) | 16.56 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint: First Occurrence of Reverse Transcription-polymerase Chain Reaction (RT-PCR) Confirmed Influenza, Due to Any Influenza Type A and/or B Virus Regardless of Antigenic Match
Description: First occurrence of RT-PCR confirmed influenza, due to any influenza Type A and/or B virus regardless of antigenic match to the influenza strains selected for the seasonal influenza vaccine, occurring at >14 days after the last vaccination and until the end of the influenza season, in association with protocol-defined influenza-like illness (ILI) symptoms
Time Frame: >14 days after last vaccination in the treatment period up to Day 181 or end of influenza season, whichever was longer (previously vaccinated subjects), or up to Day 209 or end of influenza season, whichever was longer (not previously vaccinated subjects)
Population: Full Analysis Set (FAS) Efficacy, defined as all subjects in the All Enrolled Set who were randomized, received at least one dose of study vaccination, and were evaluated for efficacy at more than 14 days after the last vaccination
Measure: Number; unit: Cases
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2856 | 2835
Cases | 104 | 173
Statistical Analysis 1: Comparison: QIVc vs Comparator; Test type: Other — The primary objective would be achieved if efficacy was demonstrated for at least one of the two primary efficacy endpoints, that is, if the interim analysis-adjusted lower limit of the two-sided confidence interval (CI) for absolute vaccine efficacy (aVE) of QIVc versus the comparator vaccine was greater than 0%; Cox Proportional Hazard = 41.26, 97.98% CI 2-sided [21.55 to 56.02]

2. Primary Outcome: Efficacy Endpoint: First Occurrence of Culture Confirmed Influenza, Due to Influenza Type A and/or B Virus Antigenically Matched by Ferret Antigenicity Testing to the Strains Selected for the Seasonal Influenza Vaccine
Description: First occurrence of culture confirmed influenza, due to influenza Type A and/or B virus antigenically matched by ferret antigenicity testing to the strains selected for the seasonal influenza vaccine, occurring at >14 days after the last vaccination and until the end of the influenza season, in association with protocol-defined ILI symptoms
Time Frame: as for outcome 1
Population: FAS Efficacy
Measure: Number; unit: Cases
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2856 | 2835
Cases | 44 | 82
Statistical Analysis 1: Comparison: QIVc vs Comparator; Test type: Other — The primary objective would be achieved if efficacy was demonstrated for at least one of the two primary efficacy endpoints, that is, if the interim analysis-adjusted lower limit of the two-sided CI for aVE of QIVc versus the comparator vaccine was greater than 0%; Cox Proportional Hazard = 46.90, 97.5% CI 2-sided [19.19 to 65.11]

3. Secondary Outcome: Efficacy Endpoint: First Occurrence of Culture Confirmed Influenza Caused by Influenza Virus Strains Antigenically Dissimilar to the Influenza Strains Selected for the Seasonal Influenza Vaccine
Description: First occurrence of culture confirmed influenza caused by influenza virus strains antigenically dissimilar to the influenza strains selected for the seasonal vaccine occurring at >14 days after the last vaccination and until the end of the influenza season, in association with protocol-defined ILI symptoms
Time Frame: as for outcome 1
Population: FAS Efficacy
Measure: Number; unit: Cases
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2856 | 2835
Cases | 20 | 43
Statistical Analysis 1: Comparison: QIVc vs Comparator; Test type: Other — The secondary efficacy objectives were not associated with any hypothesis testing; Cox Proportional Hazard = 54.49, 95% CI 2-sided [22.55 to 73.26]

4. Secondary Outcome: Efficacy Endpoint: First Occurrence of Culture Confirmed Influenza Due to Any Influenza Type A and/or Type B Virus Regardless of Antigenic Match to the Influenza Strains Selected for the Seasonal Influenza Vaccine
Description: First occurrence of culture confirmed influenza due to any influenza Type A and/or Type B virus regardless of antigenic match to the influenza strains selected for the seasonal influenza vaccine, occurring at >14 days after the last vaccination and until the end of the influenza season, in association with protocol-defined ILI symptoms
Time Frame: as for outcome 1
Population: FAS Efficacy
Measure: Number; unit: Cases
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2856 | 2835
Cases | 61 | 121
Statistical Analysis 1: Comparison: QIVc vs Comparator; Test type: Other — The secondary efficacy objectives were not associated with any hypothesis testing; Cox Proportional Hazard = 50.67, 95% CI 2-sided [32.83 to 63.77]

5. Secondary Outcome: Efficacy Endpoint: First Occurrence of RT-PCR Confirmed Moderate-to-severe Influenza Due to Any Influenza Type A and/or Type B Virus Regardless of Antigenic Match to the Influenza Strains Selected for the Seasonal Influenza Vaccine
Description: First occurrence of RT-PCR confirmed moderate-to-severe influenza due to any influenza Type A and/or Type B virus regardless of antigenic match to the influenza strains selected for the seasonal influenza vaccine, occurring at >14 days after the last vaccination and until the end of the influenza season
Time Frame: as for outcome 1
Population: FAS Efficacy
Measure: Number; unit: Cases
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2856 | 2835
Cases | 0 | 9
Statistical Analysis 1: Comparison: QIVc vs Comparator; Test type: Other — The secondary efficacy objectives were not associated with any hypothesis testing; Cox Proportional Hazard = 100 — The 2-sided 95% confidence interval was calculated with a lower limit of "not estimable" and an upper limit of 100

6. Secondary Outcome: Immunogenicity Endpoint: Prevaccination and Postvaccination Geometric Mean Titer (GMT) (HI Assay)
Description: The measures for immunogenicity are determined by a hemagglutination inhibition (HI) assay prior to first vaccination and 28 days after last vaccination for all four influenza strains
  HI = hemagglutination inhibition
  Adjusted GMTs are presented
Time Frame: Day 1 and Day 29 for previously vaccinated subjects; Day 1 and Day 57 for not previously vaccinated subjects
Population: FAS Immunogenicity, defined as all subjects in the All Enrolled Set who were randomized, received at least one study vaccination, and provided evaluable serum samples at both baseline (Day 1) and 28 days after last vaccination (Day 29/57)
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer
Groups:
- QIVc (Season 1): QIVc immunogenicity analyses (Season 1)
- Comparator (Season 1): Comparator vaccine immunogenicity analyses (Season 1)
- QIVc (Season 2): QIVc immunogenicity analyses (Season 2)
- Comparator (Season 2): Comparator vaccine immunogenicity analyses (Season 2)
- QIVc (Season 3): QIVc immunogenicity analyses (Season 3)
- Comparator (Season 3): Comparator vaccine immunogenicity analyses (Season 3)
- QIVc (Season 4): QIVc immunogenicity analyses (Season 4)
- Comparator (Season 4): Comparator vaccine immunogenicity analyses (Season 4)
- QIVc (Season 5): QIVc immunogenicity analyses (Season 5)
- Comparator (Season 5): Comparator vaccine immunogenicity analyses (Season 5)
Arm/Group | QIVc (Season 1) | Comparator (Season 1) | QIVc (Season 2) | Comparator (Season 2) | QIVc (Season 3) | Comparator (Season 3) | QIVc (Season 4) | Comparator (Season 4) | QIVc (Season 5) | Comparator (Season 5)
Number analyzed (Participants) | 112 | 108 | 107 | 111 | 111 | 112 | 87 | 85 | 108 | 108
Geometric mean titer
  A/H1N1 Day 1 HI GMT | 40.06 [21.41 to 74.97] | 44.28 [24.19 to 81.07] | 22.99 [9.52 to 55.49] | 27.50 [11.60 to 65.18] | 10.15 [4.45 to 23.13] | 8.72 [3.87 to 19.60] | 57.83 [34.41 to 97.19] | 58.00 [34.81 to 96.64] | 13.60 [1.97 to 93.97] | 13.94 [1.95 to 99.61]
  A/H1N1 Day 29/57 HI GMT | 126.39 [68.37 to 233.66] | 60.33 [33.32 to 109.21] | 60.77 [33.77 to 109.38] | 11.24 [6.32 to 20.02] | 49.38 [22.92 to 106.39] | 5.45 [2.56 to 11.58] | 149.01 [96.96 to 229.01] | 81.71 [53.55 to 124.68] | 362.71 [74.42 to 1767.89] | 60.84 [12.14 to 304.84]
  A/H3N2 Day 1 HI GMT | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | 12.21 [5.59 to 26.70] | 14.14 [6.57 to 30.41] | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | 46.38 [21.09 to 101.98] | 35.62 [16.41 to 77.30] | 82.67 [19.98 to 342.16] | 120.80 [28.47 to 512.58]
  A/H3N2 Day 29/57 HI GMT | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | 95.36 [43.91 to 207.07] | 8.79 [4.11 to 18.77] | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | 67.88 [36.64 to 125.77] | 38.85 [21.22 to 71.10] | 440.30 [127.04 to 1526.08] | 57.87 [16.29 to 205.63]
  B/Yamagata Day 1 HI GMT | 11.66 [8.26 to 16.46] | 11.53 [8.27 to 16.09] | 9.87 [6.86 to 14.22] | 8.22 [5.75 to 11.75] | 7.65 [4.25 to 13.79] | 7.54 [4.19 to 13.57] | 8.96 [6.78 to 11.84] | 9.49 [7.22 to 12.48] | 7.30 [4.19 to 12.73] | 7.35 [4.18 to 12.95]
  B/Yamagata Day 29/57 HI GMT | 18.94 [13.07 to 27.46] | 6.90 [4.82 to 9.87] | 23.65 [14.04 to 39.85] | 13.57 [8.17 to 22.53] | 13.85 [6.91 to 27.77] | 5.26 [2.63 to 10.53] | 13.80 [8.95 to 21.28] | 4.70 [3.06 to 7.22] | 53.72 [20.85 to 138.40] | 8.04 [3.07 to 21.06]
  B/Victoria Day 1 HI GMT | 7.40 [5.35 to 10.24] | 8.36 [6.11 to 11.43] | 9.37 [7.46 to 11.76] | 9.31 [7.45 to 11.63] | 8.34 [5.40 to 12.90] | 9.39 [6.12 to 14.42] | 5.82 [5.18 to 6.53] | 6.08 [5.42 to 6.82] | 7.84 [1.38 to 44.61] | 5.92 [1.01 to 34.73]
  B/Victoria Day 29/57 HI GMT | 14.97 [10.42 to 21.49] | 7.01 [4.94 to 9.95] | 16.84 [11.32 to 25.07] | 8.82 [5.97 to 13.02] | 9.54 [5.60 to 16.25] | 4.88 [2.89 to 8.26] | 23.92 [13.98 to 40.92] | 4.67 [2.73 to 7.97] | 539.53 [158.62 to 1835.19] | 45.34 [13.01 to 157.93]

7. Secondary Outcome: Immunogenicity Endpoint: Seroconversion Rates (SCR) (HI Assay)
Description: The measures for immunogenicity are determined by a HI assay prior to first vaccination and 28 days after last vaccination for all four influenza strains
  SCR is defined as the percentage of subjects with either a prevaccination HI titer <1:10 and a postvaccination HI titer ≥1:40, or a prevaccination HI titer ≥1:10 and a ≥4-fold increase in postvaccination HI titer
Time Frame: Day 1 through Day 29 for previously vaccinated subjects; Day 1 through Day 57 for not previously vaccinated subjects
Population: FAS Immunogenicity
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | QIVc (Season 1) | Comparator (Season 1) | QIVc (Season 2) | Comparator (Season 2) | QIVc (Season 3) | Comparator (Season 3) | QIVc (Season 4) | Comparator (Season 4) | QIVc (Season 5) | Comparator (Season 5)
Number analyzed (Participants) | 112 | 108 | 107 | 111 | 111 | 112 | 87 | 85 | 108 | 108
Percentage of participants
  A/H1N1 SCR HI Titer | 45.54 [36.10 to 55.22] | 12.04 [6.57 to 19.70] | 57.01 [47.08 to 66.54] | 3.60 [0.99 to 8.97] | 68.47 [58.96 to 76.96] | 2.68 [0.56 to 7.63] | 29.89 [20.54 to 40.65] | 4.71 [1.30 to 11.61] | 75.00 [65.75 to 82.83] | 12.96 [7.27 to 20.79]
  A/H3N2 SCR HI Titer | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | 70.09 [60.48 to 78.56] | 6.31 [2.57 to 12.56] | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | 44.83 [34.15 to 55.87] | 28.24 [19.00 to 39.04] | 84.26 [76.00 to 90.55] | 15.74 [9.45 to 24.00]
  B/Yamagata SCR HI Titer | 37.50 [28.53 to 47.15] | 3.70 [1.02 to 9.21] | 24.30 [16.53 to 33.54] | 6.31 [2.57 to 12.56] | 23.42 [15.91 to 32.41] | 0.90 [0.02 to 4.92] | 29.89 [20.54 to 40.65] | 1.18 [0.03 to 6.38] | 66.67 [56.95 to 75.45] | 3.70 [1.02 to 9.21]
  B/Victoria SCR HI Titer | 24.11 [16.53 to 33.10] | 2.78 [0.58 to 7.90] | 13.08 [7.34 to 20.98] | 0.90 [0.02 to 4.92] | 9.91 [5.05 to 17.04] | 0.00 [NA to NA] — Not estimable due to insufficient number of events | 42.53 [31.99 to 53.59] | 3.53 [0.73 to 9.97] | 80.56 [71.83 to 87.54] | 8.33 [3.88 to 15.23]

8. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) (HI Assay)
Description: The measures for immunogenicity are determined by a hemagglutination inhibition (HI) assay prior to first vaccination and 28 days after last vaccination for all four influenza strains
  GMR is the geometric mean of the fold increase of postvaccination HI titer over the prevaccination HI titer
  Adjusted GMRs are presented
Time Frame: Day 1 through Day 29 for previously vaccinated subjects; Day 1 through Day 57 for not previously vaccinated subjects
Population: FAS Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | QIVc (Season 1) | Comparator (Season 1) | QIVc (Season 2) | Comparator (Season 2) | QIVc (Season 3) | Comparator (Season 3) | QIVc (Season 4) | Comparator (Season 4) | QIVc (Season 5) | Comparator (Season 5)
Number analyzed (Participants) | 112 | 108 | 107 | 111 | 111 | 112 | 87 | 85 | 108 | 108
Geometric mean ratio
  A/H1N1 GMR HI Titer | 3.36 [1.69 to 6.66] | 1.53 [0.79 to 2.95] | 3.71 [2.04 to 6.73] | 0.67 [0.37 to 1.20] | 6.28 [2.91 to 13.56] | 0.70 [0.33 to 1.50] | 2.59 [1.51 to 4.45] | 1.42 [0.83 to 2.41] | 19.20 [3.61 to 102.12] | 3.20 [0.58 to 17.52]
  A/H3N2 GMR HI Titer | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | 7.43 [2.95 to 18.75] | 0.62 [0.25 to 1.54] | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | NA [NA to NA] — Not applicable due to lack of agglutination of A/H3N2 in HI assay | 1.81 [0.86 to 3.81] | 1.19 [0.57 to 2.48] | 7.14 [1.81 to 28.16] | 0.80 [0.20 to 3.24]
  B/Yamagata GMR HI Titer | 2.52 [1.75 to 3.63] | 0.92 [0.65 to 1.31] | 3.38 [2.02 to 5.67] | 1.96 [1.18 to 3.25] | 1.95 [0.91 to 4.15] | 0.75 [0.35 to 1.59] | 2.03 [1.32 to 3.13] | 0.68 [0.44 to 1.04] | 8.04 [3.12 to 20.72] | 1.20 [0.46 to 3.15]
  B/Victoria GMR HI Titer | 2.01 [1.37 to 2.96] | 0.90 [0.62 to 1.30] | 1.79 [1.15 to 2.79] | 0.94 [0.61 to 1.46] | 1.43 [0.83 to 2.44] | 0.71 [0.42 to 1.21] | 4.44 [2.62 to 7.55] | 0.85 [0.51 to 1.43] | 32.55 [8.85 to 119.71] | 2.95 [0.78 to 11.09]

9. Secondary Outcome: Immunogenicity Endpoint: Prevaccination and Postvaccination Geometric Mean Titer (GMT) (MN Assay)
Description: The measures for immunogenicity are determined by a microneutralization (MN) assay prior to first vaccination and 28 days after last vaccination for all four influenza strains
Time Frame: Day 1 and Day 29 for previously vaccinated subjects; Day 1 and Day 57 for not previously vaccinated subjects
Population: FAS Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer
Arm/Group | QIVc (Season 1) | Comparator (Season 1) | QIVc (Season 2) | Comparator (Season 2) | QIVc (Season 3) | Comparator (Season 3) | QIVc (Season 4) | Comparator (Season 4) | QIVc (Season 5) | Comparator (Season 5)
Number analyzed (Participants) | 112 | 108 | 107 | 111 | 111 | 112 | 87 | 85 | 108 | 108
Geometric mean titer
  A/H1N1 Day 1 MN GMT | 22.06 [9.53 to 51.07] | 31.10 [13.83 to 69.92] | 57.54 [18.79 to 176.16] | 55.89 [18.69 to 167.19] | 61.40 [16.51 to 228.37] | 43.43 [11.93 to 158.11] | 32.15 [19.17 to 53.90] | 35.32 [21.25 to 58.71] | 113.94 [36.64 to 354.34] | 115.49 [36.41 to 366.35]
  A/H1N1 Day 29/57 MN GMT | 329.08 [196.16 to 552.06] | 36.24 [21.97 to 59.79] | 473.15 [247.69 to 903.85] | 66.69 [35.39 to 125.71] | 459.87 [157.55 to 1342.31] | 19.32 [6.76 to 55.21] | 86.91 [58.51 to 129.11] | 46.51 [31.53 to 68.60] | 352.09 [110.01 to 1126.90] | 86.61 [26.51 to 282.92]
  A/H3N2 Day 1 MN GMT | 6.92 [4.91 to 9.76] | 6.29 [4.51 to 8.76] | 4.96 [4.19 to 5.88] | 4.80 [4.07 to 5.67] | 7.02 [3.18 to 15.51] | 8.33 [3.82 to 18.16] | 17.70 [10.34 to 30.31] | 15.77 [9.29 to 26.76] | 26.08 [7.79 to 87.37] | 25.98 [7.59 to 88.87]
  A/H3N2 Day 29/57 MN GMT | 27.55 [18.70 to 40.58] | 10.95 [7.52 to 15.94] | 12.04 [7.60 to 19.08] | 5.31 [3.38 to 8.34] | 57.93 [28.43 to 118.06] | 10.49 [5.21 to 21.09] | 35.99 [18.52 to 69.94] | 14.78 [7.70 to 28.34] | 139.97 [41.52 to 471.84] | 30.22 [8.78 to 104.08]
  B/Yamagata Day 1 MN GMT | 76.91 [53.50 to 110.55] | 66.14 [46.60 to 93.87] | 65.25 [35.87 to 118.70] | 60.03 [33.41 to 107.86] | 15.33 [7.73 to 30.41] | 15.26 [7.78 to 29.93] | 53.41 [32.42 to 88.00] | 54.11 [33.12 to 88.41] | 51.81 [23.27 to 115.35] | 45.20 [20.02 to 102.06]
  B/Yamagata Day 29/57 MN GMT | 278.89 [202.31 to 384.46] | 88.67 [65.06 to 120.84] | 283.42 [183.07 to 438.79] | 126.59 [82.43 to 194.41] | 55.17 [27.19 to 111.92] | 19.24 [9.59 to 38.59] | 84.60 [55.74 to 128.38] | 52.11 [34.57 to 78.55] | 169.24 [75.01 to 381.86] | 49.34 [21.58 to 112.85]
  B/Victoria Day 1 MN GMT | 6.07 [4.82 to 7.65] | 6.64 [5.31 to 8.30] | 4.99 [4.16 to 5.99] | 5.18 [4.33 to 6.18] | 9.09 [4.80 to 17.24] | 10.71 [5.71 to 20.09] | 8.79 [6.40 to 12.07] | 7.72 [5.66 to 10.55] | 15.97 [2.53 to 100.98] | 12.20 [1.87 to 79.68]
  B/Victoria Day 29/57 MN GMT | 14.23 [10.95 to 18.51] | 7.00 [5.44 to 9.02] | 5.29 [4.03 to 6.92] | 5.26 [4.04 to 6.85] | 26.81 [14.06 to 51.12] | 9.65 [5.12 to 18.20] | 121.02 [59.56 to 245.87] | 5.99 [2.99 to 11.97] | 938.65 [230.67 to 3819.51] | 39.32 [9.41 to 164.32]

10. Secondary Outcome: Immunogenicity Endpoint: Seroconversion Rates (SCR) (MN Assay)
Description: The measures for immunogenicity are determined by a MN assay prior to first vaccination and 28 days after last vaccination for all four influenza strains
  SCR is defined as the percentage of subjects with either a prevaccination MN titer <1:10 and a postvaccination MN titer ≥1:40, or a prevaccination MN titer ≥1:10 and a ≥4-fold increase in postvaccination MN titer
Time Frame: Day 1 through Day 29 for previously vaccinated subjects; Day 1 through Day 57 for not previously vaccinated subjects
Population: FAS Immunogenicity
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | QIVc (Season 1) | Comparator (Season 1) | QIVc (Season 2) | Comparator (Season 2) | QIVc (Season 3) | Comparator (Season 3) | QIVc (Season 4) | Comparator (Season 4) | QIVc (Season 5) | Comparator (Season 5)
Number analyzed (Participants) | 112 | 108 | 107 | 111 | 111 | 112 | 87 | 85 | 108 | 108
Percentage of participants
  A/H1N1 SCR (%) MN Titer | 73.21 [64.02 to 81.14] | 2.78 [0.58 to 7.90] | 74.77 [65.45 to 82.67] | 4.50 [1.48 to 10.20] | 87.39 [79.74 to 92.93] | 4.46 [1.47 to 10.11] | 32.18 [22.56 to 43.06] | 7.06 [2.63 to 14.73] | 68.52 [58.88 to 77.12] | 15.74 [9.45 to 24.00]
  A/H3N2 SCR (%) MN Titer | 38.39 [29.36 to 48.06] | 4.63 [1.52 to 10.47] | 20.56 [13.36 to 29.46] | 1.80 [0.22 to 6.36] | 57.66 [47.92 to 66.98] | 1.79 [0.22 to 6.30] | 33.33 [23.58 to 44.25] | 10.59 [4.96 to 19.15] | 71.30 [61.80 to 79.59] | 15.74 [9.45 to 24.00]
  B/Yamagata SCR (%) MN Titer | 46.43 [36.95 to 56.10] | 0.93 [0.02 to 5.05] | 30.84 [22.27 to 40.50] | 3.60 [0.99 to 8.97] | 36.94 [27.97 to 46.62] | 4.46 [1.47 to 10.11] | 19.54 [11.81 to 29.43] | 4.71 [1.30 to 11.61] | 54.63 [44.76 to 64.24] | 7.41 [3.25 to 14.07]
  B/Victoria SCR (%) MN Titer | 20.54 [13.49 to 29.20] | 0.93 [0.02 to 5.05] | 0.93 [0.02 to 5.10] | 2.70 [0.56 to 7.70] | 25.23 [17.46 to 34.35] | 0.89 [0.02 to 4.87] | 87.36 [78.50 to 93.52] | 7.06 [2.63 to 14.73] | 94.44 [88.30 to 97.93] | 9.26 [4.53 to 16.37]

11. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) (MN Assay)
Description: The measures for immunogenicity are determined by a MN assay prior to first vaccination and 28 days after last vaccination for all four influenza strains GMR is the geometric mean of the fold increase of post-vaccination MN titer over the pre-vaccination MN titer
Time Frame: Day 1 through Day 29 for previously vaccinated subjects; Day 1 through Day 57 for not previously vaccinated subjects
Population: FAS Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | QIVc (Season 1) | Comparator (Season 1) | QIVc (Season 2) | Comparator (Season 2) | QIVc (Season 3) | Comparator (Season 3) | QIVc (Season 4) | Comparator (Season 4) | QIVc (Season 5) | Comparator (Season 5)
Number analyzed (Participants) | 112 | 108 | 107 | 111 | 111 | 112 | 87 | 85 | 108 | 108
Geometric mean ratio
  A/H1N1 GMR MN Titer | 16.16 [9.52 to 27.45] | 1.70 [1.02 to 2.83] | 8.12 [4.19 to 15.75] | 1.15 [0.60 to 2.20] | 17.55 [5.72 to 53.86] | 0.81 [0.27 to 2.44] | 2.37 [1.54 to 3.67] | 1.23 [0.80 to 1.88] | 3.47 [1.07 to 11.24] | 0.85 [0.26 to 2.81]
  A/H3N2 GMR MN Titer | 3.28 [2.23 to 4.84] | 1.32 [0.91 to 1.92] | 2.14 [1.35 to 3.40] | 0.93 [0.59 to 1.46] | 5.92 [2.79 to 12.56] | 1.01 [0.48 to 2.13] | 2.74 [1.39 to 5.38] | 1.16 [0.60 to 2.26] | 4.40 [1.30 to 14.88] | 0.95 [0.27 to 3.28]
  B/Yamagata GMR MN Titer | 3.93 [2.81 to 5.49] | 1.30 [0.94 to 1.79] | 3.05 [1.95 to 4.75] | 1.38 [0.89 to 2.13] | 3.15 [1.47 to 6.71] | 1.10 [0.52 to 2.32] | 1.82 [1.15 to 2.88] | 1.11 [0.71 to 1.75] | 3.81 [1.56 to 9.33] | 1.19 [0.48 to 2.95]
  B/Victoria GMR MN Titer | 2.17 [1.67 to 2.82] | 1.07 [0.83 to 1.37] | 1.04 [0.77 to 1.40] | 1.01 [0.75 to 1.35] | 2.74 [1.37 to 5.47] | 0.92 [0.47 to 1.83] | 16.90 [8.36 to 34.19] | 0.86 [0.43 to 1.72] | 31.51 [7.19 to 138.05] | 1.42 [0.31 to 6.37]

12. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Solicited Local and Systemic Adverse Events (AEs)
Description: Percentage of subjects with solicited local and systemic AEs assessed for 7 days following each vaccination in the QIVc group and in the comparator group
Time Frame: 7 days following each vaccination in the treatment period, ie, Day 1 to Day 7 for previously vaccinated subjects and Day 1 to Day 7 and Day 29 to Day 35 for not previously vaccinated subjects
Population: Solicited Safety Set, defined as all subjects in the All Exposed Set with any solicited AE data indicating the occurrence or lack of occurrence of solicited AEs, ie, a subject does not have to have any solicited AEs to be included in this population
Measure: Number; unit: Percentage of participants
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2813 | 2790
Percentage of participants
  Solicited AEs | 55.8 | 60.8
  Solicited Local AEs | 32.3 | 40.4
  Solicited Systemic AEs | 40.9 | 42.5
  Analgesic/Antipyretic Use | 14.5 | 15.0

13. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Unsolicited AEs
Description: Percentage of subjects with any unsolicited AEs assessed in the QIVc group and in the comparator group until 28 days after each vaccination
Time Frame: 28 days after each vaccination in the treatment period, ie, Day 1 to Day 29 for previously vaccinated subjects and Day 1 to Day 57 for not previously vaccinated subjects
Population: Unsolicited Safety Set, defined as all subjects in the All Exposed Set with unsolicited AE data
Measure: Number; unit: Percentage of participants
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2856 | 2841
Percentage of participants
  Any AE | 42.5 | 45.4
  Any related AE | 4.2 | 3.6

14. Secondary Outcome: Safety Endpoint: Percentage of Subjects With SAEs, NOCDs, AEs Leading to Withdrawal From the Study or Vaccination
Description: Percentage of subjects with serious adverse events (SAEs), new onset of chronic disease (NOCD), AEs leading to withdrawal from the study or vaccination, and all medications associated with these events in the QIVc group and in the comparator group
  Note: The time frame for assessment of these AEs was Day 1 through Study Completion as indicated below. Subjects aged 6 months through 11 months at enrollment in countries without NeisVac-C vaccine marketing authorization had an additional study visit 28 days later (ie, Day 237).
Time Frame: Day 1 through Study Completion, ie, Day 1 to Day 181 or end of influenza season, whichever was longer, for previously vaccinated subjects and Day 1 to Day 209 or end of influenza season, whichever was longer, for not previously vaccinated subjects
Population: Unsolicited Safety Set
Measure: Number; unit: Percentage of participants
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2856 | 2841
Percentage of participants
  SAE | 2.2 | 3.0
  Related SAE | 0 | 0.04
  NOCD | 0.7 | 0.4
  AE leading to study withdrawal | 0 | 0
  AE leading to study vaccine withdrawal | 0 | 0.1

15. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Medically-attended AEs
Description: Percentage of subjects with medically-attended AEs within 30 days after ILI onset in the QIVc group and in the comparator group
Time Frame: If a subject experienced an ILI during approximately 8 months of study participation, medically-attended AEs were collected for the 30-day period after onset of the ILI (defined as the first day that a subject meets the criteria for protocol-defined ILI)
Population: Unsolicited Safety Set
Measure: Number; unit: Percentage of participants
Arm/Group | QIVc | Comparator
Number analyzed (Participants) | 2856 | 2841
Percentage of participants | 28.9 | 32.6

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: Day 1 through Study Completion, ie, Day 1 to Day 181/end of influenza season for previously vaccinated subjects and Day 1 to Day 209/end of influenza season for not previously vaccinated subjects Solicited AEs: 7 days following each vaccination in the treatment period, ie, Day 1 to Day 7 for previously vaccinated subjects and Day 1 to Day 7 and Day 29 to Day 35 for not previously vaccinated subjects
Description: Number and percentage of subjects with SAEs and other AEs (ie, nonserious unsolicited AEs and solicited AEs)
  All-cause mortality, SAEs, and nonserious AEs are reported for the Unsolicited Safety Set; solicited AEs are reported for the Solicited Safety Set
  None of the deaths in the study were assessed as related to study vaccine
  All AEs are reported according to the intervention subjects received in the treatment period
Arm/Group | QIVc | Comparator
All-Cause Mortality (participants affected / at risk) | 1/2856 | 2/2841
Serious Adverse Events (participants affected / at risk) | 64/2856 | 84/2841
Other Adverse Events (participants affected / at risk) | 2050/2856 | 2126/2841
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QIVc (N=2856) | Comparator (N=2841)
Pneumonia (Infections and infestations) | 15 | 24
Gastroenteritis (Infections and infestations) | 8 | 12
Dengue fever (Infections and infestations) | 6 | 7
Viral infection (Infections and infestations) | 4 | 0
Influenza (Infections and infestations) | 3 | 6
Bronchiolitis (Infections and infestations) | 2 | 3
Otitis media acute (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 2 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 2 | 0
Typhoid fever (Infections and infestations) | 2 | 1
Abscess neck (Infections and infestations) | 1 | 0
Amoebic dysentery (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 3
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1
Norovirus infection (Infections and infestations) | 1 | 2
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Abscess limb (Infections and infestations) | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 2
Amoebiasis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis adenovirus (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 3
Febrile convulsion (Nervous system disorders) | 5 | 3
Seizure (Nervous system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Kawasaki's disease (Vascular disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QIVc (N=2856) | Comparator (N=2841)
Upper respiratory tract infection (Infections and infestations) | 576 | 634
Rhinitis (Infections and infestations) | 282 | 290
Nasopharyngitis (Infections and infestations) | 255 | 255
Respiratory tract infection (Infections and infestations) | 162 | 158
Injection site pain (General disorders) | 816 | 889
Injection site erythema (General disorders) | 717 | 884
Injection site induration (General disorders) | 464 | 730
Injection site bruising (General disorders) | 303 | 339
Pyrexia (General disorders) | 307 | 307
Irritability (Psychiatric disorders) | 659 | 706
Eating disorder (Psychiatric disorders) | 447 | 455
Somnolence (Nervous system disorders) | 514 | 522
Diarrhoea (Gastrointestinal disorders) | 372 | 372
Vomiting (Gastrointestinal disorders) | 188 | 207

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication by Institution or Investigator shall not be made before the first multicenter publication of the entire study results. Seqirus must be notified of any intent to publish data collected from the study and prior approval from Seqirus must be obtained prior to submission for publication.

DOCUMENTS (2):
  • Study Protocol (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT03932682/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT03932682/SAP_001.pdf